CLINICAL TRIAL: NCT04658680
Title: Can BCG Vaccination at First Health-facility Contact Reduce Early Infant Mortality? A Cluster Randomised Trial
Brief Title: Can BCG Vaccination at First Health-facility Contact Reduce Early Infant Mortality?
Acronym: CS-BCG
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 062/CNES/INASA/2020
Record Dates: First submitted 2020-11-19; First posted 2020-12-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Infant Mortality; BCG
Keywords: Non-specific effects of vaccines
MeSH Terms: conditions — Infant Death

STUDY DESIGN:
Intervention Model Description: All participants live in the catchment areas of one of 23 HFs. The HFs will be randomized to either BCG vaccination per usual practice or to extended BCG availability. The randomization of HFs will be crossed over after 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG available at first health facility contact (Experimental): Infants living in catchment areas of HFs randomized to opening of BCG vial if just 1 eligible child is present.
  Interventions: Drug: BCG vaccination at first health facility contact
- Usual availability of BCG at health facilities (No Intervention): Infants living in catchment areas of HFs randomized to BCG availability according to the per usual restricted vial opening policy aiming at reducing vaccine wastage. This entails that BCG vaccination is commonly only available on specific predefined days where a BCG vial will only be opened if several children are present.

INTERVENTIONS:
Drug: BCG vaccination at first health facility contact — Intradermal injection at first health facility contact: 0.05 ml dose Mycobacterium bovis BCG live attenuated vaccine in the left deltoid region.
  The strain supplied by the national vaccination programme is provided through UNICEF. Different strains are used interchangeably. The additional BCG vaccines provided through this study will be procured by the Bandim Health Project. Vaccines will be from the WHO list of prequalified vaccines and the same strain will be used in intervention and control health centres.
  Arms: BCG available at first health facility contact

SUMMARY:
Bacillus Calmette-Guérin (BCG) vaccination is recommended at birth to protect against tuberculosis (TB) in countries with high TB burden. BCG is supplied in multidose vials with limited durability after reconstitution. In Guinea-Bissau, this has led to a practice of only opening a BCG vial at specific days, and only if sufficient children are present. Therefore, BCG vaccination is frequently delayed. Accumulating evidence indicates that BCG has beneficial effects on survival beyond the specific protection against tuberculosis, so called non-specific effects (NSEs).

The hypothesis of this study is that increasing the availability of BCG and vaccinating children at the first health-facility contact can reduce early infant non-accidental mortality by 25%.

In a cluster-randomised crossover trial, 23 health facilities (HFs) in three rural regions in Guinea-Bissau will be randomised to either continue with current practice (typically BCG vaccination once a week if a sufficient number of children are present for vaccination); or to offer additional BCG vaccines to make BCG available every day and open a vial of BCG if there is just one eligible child present. All children born in the three regions and registered during the study period, will be eligible for inclusion into the trial 1 day after birth. If consent is given by the mother, the child will be followed until day 42 after birth, when other vaccines are scheduled to be given. The primary outcome will be non-accidental mortality, secondary outcomes are non-accidental hospital admissions, non-accidental neonatal mortality and cost-effectiveness of making BCG available at the first health-facility contact.

DETAILED DESCRIPTION:
Background:

The World Health Organization (WHO) recommends Bacillus Calmette-Guérin (BCG) vaccination at birth to protect against TB in countries with high TB burden. Though the BCG vaccine is scheduled at birth, the vaccine is often given with delay, also among children born in Health Facilities (HFs), where it should be possible to obtain the vaccine. In 2010 in rural Guinea-Bissau, only 38% of children received BCG within the first month of life. BCG is supplied in 20-dose vials and unused doses must be discarded 6 hours after reconstitution. This has led to a local practice of not opening a BCG vial unless sufficient eligible children are present for vaccination. Moreover, the HFs seek to assemble larger groups of children eligible for BCG at specific days. Our observations from the field indicate that even on these days, vials may not be opened if the number of children is too low. Similar practises have been demonstrated in other low-income countries, but this practice is not in line with WHO recommendations, which emphasise that multi-dose vials should be opened and used to vaccinate one child despite any wastage.

In 2012, an estimated 73% of all neonatal deaths occurred within the first week of life. Several studies have suggested that BCG vaccination is associated with survival benefits early in life: In three randomised trials from Guinea-Bissau, BCG-at-birth was associated with a 38% lower neonatal mortality and marked reductions already 3 days after vaccination. A WHO-commissioned review and meta-analysis conducted in 2014 including five clinical trials indicated that BCG-vaccinated children had a relative risk of mortality at 0.70 (95% confidence interval 0.49-1.01) compared with BCG-unvaccinated children. Two randomised trials from India, both published after the review was conducted, found no effect of BCG at birth on neonatal mortality. In both India and Guinea-Bissau, all trials were conducted among low birth weight (LBW) children and primary outcome was neonatal mortality. In Guinea-Bissau, BCG-Denmark was used in all trials, whereas BCG-Russia was used in the trials from India. Strain of BCG has been suggested as a possible reason for the discrepancy between the trials in India, and the trials in Guinea-Bissau.

Therefore, early BCG vaccination may be important, not only for protection against tuberculosis, but also for the impact on survival.

Hypothesis:

Increasing the availability of BCG and vaccinating children at the first health-facility contact can reduce early infant mortality due to other causes than accidents by 25%.

Methods:

This study will be a cluster randomized trial of increased BCG availability at the 23 HFs in three rural regions (Oio, Biombo and Farim) in Guinea-Bissau. In half of the HFs, BCG will be provided as per current practice (typically once a week if a sufficient number of children are present for vaccination); in the remaining HFs, additional BCG vaccines will be supplied to make BCG available every day and opening a vial of BCG if there is just one eligible child present. In collaboration with the national vaccination programme, the investigators will ensure that the same strain of WHO-prequalified BCG vaccines will be used at the same time in both the control and intervention arm of the study. The allocation of centres will be crossed over after 12 months and inclusion of participants will carry on for another 12 months. Pregnancies, births and deaths will be monitored through two different levels of surveillance:

Level 1 - Bandim Health Project's (BHPs) rural Health and Demographic Surveillance System (HDSS). The BHP teams survey women of fertile age and children below the age of 5 years in randomly selected village clusters in all health regions across the country, which involves 40 village clusters distributed across the three regions included in this study. Through this system, it is possible to monitor pregnancies, births, vaccinations and child health.

Level 2 - Reinforced community health worker monitoring. In all villages in Guinea-Bissau, community health workers (CHWs) monitor births and deaths through a national monitoring system. The CHWs report aggregated data on pregnancies, number of births and neonatal deaths (in two categories: 0-7 days, 8-28 days) in their capture area to the local health centre at monthly meetings. This data collection will be reinforced by supervision and further data collection from BHP supervisors covering each health centre area. The CHWs will receive a visit every 1-2 months from a supervisor.

All children registered during pregnancy in Oio, Biombo or Farim enter the trial cohort 1 day after birth. A pregnancy can be registered in more than one village, but the child will only enter the trial if the mother gave birth in the village or the nearby health facility, and then was discharged to the village where the pregnancy was registered.

For all registered deaths, a specially trained field worker will visit the household of the deceased child to conduct a verbal autopsy.

Prior to study start, all 23 HFs in the three regions will be visited by a team from BHP. During these visits, refresher training on vaccination technique and assessment of lymph glands will be conducted. The training will include general information on the BCG vaccine, information on reconstitution and durability of the vaccines, how to check that the vials have not been damaged by heat and information on adverse events. During the trial, the HFs will be visited regularly by a nurse from BHP, who will observe and supervise the vaccination sessions for vaccination technique, attention to registration of adverse event, used strain of vaccinations, registration of cold chain and state of vaccine stock.

Statistical analyses:

The primary outcome will be non-accidental mortality rate between 1 day after birth and 42 days after birth, where other vaccines are scheduled to be given. 22,800 infants are expected to be included in the study during the two-year study period. With a baseline mortality of 2.5% (varying between 1.5 and 3.5% by HF) this sample size should result in 88% power to demonstrate an effect if the true mortality reduction is assumed to be 25% (power simulations based on a logistic regression with Generalised Estimating Equation (GEE)-based correction for village cluster). Secondary outcomes are non-accidental hospital admissions, non-accidental neonatal mortality and cost-effectiveness of making BCG available at the first health-facility contact. The effect of making BCG available at the first HF contact will be analysed in logistic regression models with GEE-based correction for village cluster.

ELIGIBILITY:
Inclusion Criteria:

* All children registered during pregnancy in Oio, Biombo or Farim by CHWs or the BHP HDSS

Exclusion Criteria:

* Children, who have died within 1 day after birth
* Children born outside Oio, Biombo and Farim health regions

Ages: 1 Day to 42 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22800 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Odds ratio of non-accidental early infant mortality | From 1 day after birth to 42 days after birth
  The primary analysis of early infant non-accidental mortality will be assessed in an intention-to-treat (TT) analysis. Logistic regression models with generalised estimating equation (GEE) correction for village cluster will be used.
  Furthermore, an assessment of whether the effect of the intervention on the primary outcome is modified by the following potential effect modifiers, will be carried out: Sex, maternal BCG scar (yes/no), season of birth (dry/rainy), strain of BCG.

SECONDARY OUTCOMES:
Odds ratio of non-accidental neonatal mortality | From 1 day after birth to 28 days after birth
  Assessment of the effect of BCG availability on the village cluster level non-accidental neonatal mortality based on CHW registration.
Odds ratio of severe morbidity | From 1 day after birth to 42 days after birth
  Non-accidental hospital admissions (defined as overnight hospitalisations or arrival at the hospital and death within the first day) defined by the following potential effect modifiers: sex, maternal BCG scar (yes/no), season of birth (dry/rainy), strain of BCG.
Incremental cost-effectiveness ratio per death averted by making BCG available at the first health facility contact | From 1 day after birth to 42 days after birth
  A cost-effectiveness analysis estimating the incremental costs per death averted by making BCG available at the first health facility contact will be undertaken. Incremental costs will be assessed by contrasting the costs of BCG vaccine provision in the present programme and in a scenario with BCG available at the first health-facility contact as tested in the trial. The costs/savings associated with different rates of consultations and admissions will also be taken into account. This analysis will only be carried out, if the analysis of the primary outcome shows that increasing availability of BCG reduces early infant mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ane B Fisker, MD, PhD, Principal Investigator — Bandim Health Project and University of Southern Denmark; Andreas M Jensen, MSc, Principal Investigator — Bandim Health Project and University of Southern Denmark; Julie O Vedel, MD, Principal Investigator — Bandim Health Project and University of Southern Denmark; Sanne M Thysen, MD, PhD, Study Director — Bandim Health Project and Center for Clinical Research and Prevention, Hospital of Bispebjerg and Frederiksberg; Christine S Benn, MD,PhD,DMSc, Study Director — Bandim Health Project and University of Southern Denmark; Peter Aaby, DMSc, Study Director — Bandim Health Project; Aksel Jensen, MSc, PhD, Study Director — Department of Public Health, University of Copenhagen
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected as part of the study will be available upon request in anonymized form.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After conclusion of the study period.
Access Criteria: Data will be available on a collaborative basis. Please contact a.fisker@health.sdu.dk

REFERENCES:
- [Background] World Health Organization. BCG vaccine: WHO position paper, February 2018 - Recommendations. Vaccine. 2018 Jun 7;36(24):3408-3410. doi: 10.1016/j.vaccine.2018.03.009. Epub 2018 Mar 30. PMID 29609965
- [Background] Thysen SM, Byberg S, Pedersen M, Rodrigues A, Ravn H, Martins C, Benn CS, Aaby P, Fisker AB. BCG coverage and barriers to BCG vaccination in Guinea-Bissau: an observational study. BMC Public Health. 2014 Oct 4;14:1037. doi: 10.1186/1471-2458-14-1037. PMID 25282475
- [Background] Kagone M, Ye M, Nebie E, Sie A, Schoeps A, Becher H, Muller O, Fisker AB. Vaccination coverage and factors associated with adherence to the vaccination schedule in young children of a rural area in Burkina Faso. Glob Health Action. 2017;10(1):1399749. doi: 10.1080/16549716.2017.1399749. PMID 29185899
- [Background] Wallace AS, Willis F, Nwaze E, Dieng B, Sipilanyambe N, Daniels D, Abanida E, Gasasira A, Mahmud M, Ryman TK. Vaccine wastage in Nigeria: An assessment of wastage rates and related vaccinator knowledge, attitudes and practices. Vaccine. 2017 Dec 4;35(48 Pt B):6751-6758. doi: 10.1016/j.vaccine.2017.09.082. Epub 2017 Oct 21. PMID 29066189
- [Background] Mutua, M.K., et al. Analysis of Fully Immunized Child (FIC), Associated Factors, Outcomes, and Impact Using Routinely Population Cohort Data 2001-2014. Report by the INDEPTH Network as a collaboration with GAVI 2015 18th April 2020 ]; Available from: http://www.indepth-network.org/sites/default/files/content/project_pages/files/Fully%20Immunized%20Child%20Report%20and%20Appendices.pdf.
- [Background] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Roth A, Jensen H, Garly ML, Djana Q, Martins CL, Sodemann M, Rodrigues A, Aaby P. Low birth weight infants and Calmette-Guerin bacillus vaccination at birth: community study from Guinea-Bissau. Pediatr Infect Dis J. 2004 Jun;23(6):544-50. doi: 10.1097/01.inf.0000129693.81082.a0. PMID 15194836
- [Background] Biering-Sorensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, Schaltz-Buchholzer F, Jorgensen ASP, Rodrigues A, Fisker AB, Benn CS. Early BCG-Denmark and Neonatal Mortality Among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis. 2017 Oct 1;65(7):1183-1190. doi: 10.1093/cid/cix525. PMID 29579158
- [Background] Schaltz-Buchholzer F, Biering-Sorensen S, Lund N, Monteiro I, Umbasse P, Fisker AB, Andersen A, Rodrigues A, Aaby P, Benn CS. Early BCG Vaccination, Hospitalizations, and Hospital Deaths: Analysis of a Secondary Outcome in 3 Randomized Trials from Guinea-Bissau. J Infect Dis. 2019 Jan 29;219(4):624-632. doi: 10.1093/infdis/jiy544. PMID 30239767
- [Background] Jayaraman K, Adhisivam B, Nallasivan S, Krishnan RG, Kamalarathnam C, Bharathi M, McSharry B, Namachivayam SP, Shann F, Boopalan SI, David P, Bhat BV. Two Randomized Trials of the Effect of the Russian Strain of Bacillus Calmette-Guerin Alone or With Oral Polio Vaccine on Neonatal Mortality in Infants Weighing <2000 g in India. Pediatr Infect Dis J. 2019 Feb;38(2):198-202. doi: 10.1097/INF.0000000000002198. PMID 30256314
- [Background] Curtis N. BCG Vaccination and All-Cause Neonatal Mortality. Pediatr Infect Dis J. 2019 Feb;38(2):195-197. doi: 10.1097/INF.0000000000002230. No abstract available. PMID 30640189
- [Background] Thysen SM, Benn CS, Gomes VF, Rudolf F, Wejse C, Roth A, Kallestrup P, Aaby P, Fisker A. Neonatal BCG vaccination and child survival in TB-exposed and TB-unexposed children: a prospective cohort study. BMJ Open. 2020 Feb 28;10(2):e035595. doi: 10.1136/bmjopen-2019-035595. PMID 32114478
- [Derived] Thysen SM, Moller Jensen A, Vedel JO, da Silva Borges I, Aaby P, Jensen AKG, Benn CS, Fisker AB. Can BCG vaccination at first health-facility contact reduce early infant mortality? Study protocol for a cluster-randomised trial (CS-BCG). BMJ Open. 2022 Nov 21;12(11):e063872. doi: 10.1136/bmjopen-2022-063872. PMID 36410811